CLINICAL TRIAL: NCT04837391
Title: Evaluation of the Relationship Between Postoperative Cognitive Dysfunction and Brain Injury Biomarkers In Geriatric Urologic Oncology Patients
Brief Title: Postoperative Cognitive Dysfunction in Elderly Urologic Oncology Patients (POCD)
Acronym: POCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Other Study IDs: 2019/1555
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium; Frailty
Keywords: postoperative cognitive dysfunction; frailty; S 100β; NSE; IL-6; HMGB-1 protein; NIRS; geriatric anesthesia
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium; Frailty | interventions — Spectroscopy, Near-Infrared; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected from study participants after anesthesia induction and after the end of the operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urologic oncology surgery in elderly: Elective urologic oncology surgeries such as radical nephrectomy, radical cystectomy, radical prostatectomy in older than 65 years
  Interventions: Device: Near Infrared Spectroscopy (NIRS); Diagnostic Test: Blood sample; Diagnostic Test: Addenbrooke Cognitive Examination III (ACE-III); Diagnostic Test: Confusion Assessment Method

INTERVENTIONS:
Device: Near Infrared Spectroscopy (NIRS) — Patients are monitored by near infrared spectroscopy before anesthesia induction until end of the operation. Graphical presentation of cerebral oxygenation during surgery evaluated by INVOS Analytics Tool Version 1.2.
  Other Names: INVOS Cerebral Oximeter 5100C (Covidien Dublin, Ireland)
Diagnostic Test: Blood sample — Blood samples are obtained before and after surgery. S-100, Neuron specific enolase (NSE), Interleukin-6 (IL-6), High Mobility Group Box Protein (HMGB-1) are going to be studied by ELISA method after data collection process end.
Diagnostic Test: Addenbrooke Cognitive Examination III (ACE-III) — ACE-III is administered to study participants one day before surgery, 1 week after surgery, and three months after surgery to diagnose postoperative cognitive dysfunction.
Diagnostic Test: Confusion Assessment Method — Confusion Assessment Method is administered to study participants in postoperative recovery room to diagnose postoperative delirium.

SUMMARY:
Postoperative cognitive changes are more common in elderly patients, which can result in poor quality of life, loss of workforce, disability, early retirement, physical-social dependence, increased health care cost and premature mortality. Postoperative cognitive complications are also quite common in extensive oncological surgeries. In this study, our aim is to evaluate the relationship between the development of postoperative cognitive dysfunction (POCD) in geriatric urologic oncology patients with brain injury and inflammatory markers [S100 β, neuron specific enolase (NSE), interleukin 6 (IL-6) and high mobility group box-1 (HMGB-1 protein)].

DETAILED DESCRIPTION:
The incidence of POCD changes by age group, type of surgery, testing neuropsychological tests, timing of tests, and the method used for diagnosis. In non-cardiac surgery over the age of 60; the incidence of POCD was 26% in the postoperative 1st week and 10% in the postoperative 3rd month. Although old age is an important risk factor, POCD incidence of up to 36.6% has been reported in a younger period. Major cancer surgery is an important risk factor for development of POCD.

Numerous biomarkers such as; S100β, NSE, Human IL-6, HMGB-1 protein; have been evaluated in studies to determine the diagnosis, prognosis, stage and treatment of POCD.

In this study, our aim is to evaluate the relationship between the development of postoperative cognitive dysfunction (POCD) in geriatric urologic oncology patients with brain injury and inflammatory markers. (S100β, NSE, Human IL-6 and HMGB-1 protein).The hypothesis of our study is that postoperative brain injury and inflammatory markers (S100β, NSE, Human IL-6 and HMGB-1 protein) will be higher in patients who develop POCD compared to patients who do not develop POCD in geriatric urologic oncology surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 65 who are planned to undergo major urooncological surgery.

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Patients with severe hearing-vision problems.
* Patients with serious neurological-psychiatric disorders.
* Patients with language barrier.
* Patients with missing in any interventions.
* Patients with blood samples that are not suitable for the ELISA.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over the age of 65 who are planned to undergo major urooncological surgery (radical nephrectomy, radical prostatectomy and radical cystectomy) as of April 21, 2020 at the Istanbul University Hospital are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-05-21 (Estimated); Study Completion 2021-07-21 (Estimated)

PRIMARY OUTCOMES:
Addenbrooke cognitive examination at the day before surgery. | The day before surgery.
  Test score is between 0-100. 100 is the best point and 0 is the worst point in the test. The test has five cognitive domains including attention, memory, language, visuospatial function, and verbal fluency. Patients who score less than 88 in preoperative tests will be diagnosed with mild cognitive impairment.
Addenbrooke cognitive examination at seventh day after surgery. | The seventh day after surgery.
  POCD is diagnosed by 1 standard deviation decrease from the preoperative test scores.
Addenbrooke cognitive examination at third months after surgery. | The third months after surgery.
  POCD is diagnosed by 1 standard deviation decrease from the preoperative test scores.
S 100β (pg/mL) | Change from baseline serum concentration of S 100 β at 6 hours
  Blood S 100β concentration is determined by an enzyme-linked immunosorbent assay kit.
High Mobility Group Box1 Protein (HMGB1) (ng/mL) | Change from baseline serum concentration of HMGB1 at 6 hours
  HMGB1 concentration is determined by an enzyme-linked immunosorbent assay kit.
Human Neuron Specific Enolase (h-NSE) (ng/mL) | Change from baseline serum concentration of h-NSE at 6 hours
  h-NSE concentration is determined by an enzyme-linked immunosorbent assay kit.
Interleukine-6 (IL-6) (pg/mL) | Change from baseline serum concentration of IL-6 at 6 hours
  Blood IL-6 concentration is determined by an enzyme-linked immunosorbent assay kit.

SECONDARY OUTCOMES:
Postoperative delirium | Up to postoperative day one
  Postoperative delirium is diagnosed by confusion assessment method.
Cerebral oxygenation | During surgery
  Cerebral hypoxia is defined as reduction of regional oxygen saturation by 10 % from baseline before surgery.
Overall postoperative complications | Up to postoperative three months.
  Stroke, transient ischemic attack, arrhythmia, heart failure, myocardial injury, respiratory failure, pneumonia, ileus, acute kidney injury, prolonged length of stay, mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, Assoc. Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yanagisawa R, Tanaka M, Yashima F, Arai T, Kohno T, Shimizu H, Fukuda K, Naganuma T, Mizutani K, Araki M, Tada N, Yamanaka F, Shirai S, Tabata M, Ueno H, Takagi K, Higashimori A, Watanabe Y, Yamamoto M, Hayashida K. Frequency and Consequences of Cognitive Impairmentin Patients Underwent Transcatheter Aortic Valve Implantation. Am J Cardiol. 2018 Sep 1;122(5):844-850. doi: 10.1016/j.amjcard.2018.05.026. Epub 2018 Jun 2. PMID 30072128
- [Background] Rundshagen I. Postoperative cognitive dysfunction. Dtsch Arztebl Int. 2014 Feb 21;111(8):119-25. doi: 10.3238/arztebl.2014.0119. PMID 24622758
- [Background] Plas M, Rotteveel E, Izaks GJ, Spikman JM, van der Wal-Huisman H, van Etten B, Absalom AR, Mourits MJE, de Bock GH, van Leeuwen BL. Cognitive decline after major oncological surgery in the elderly. Eur J Cancer. 2017 Nov;86:394-402. doi: 10.1016/j.ejca.2017.09.024. Epub 2017 Nov 5. PMID 29100194
- [Background] Kapoor I, Prabhakar H, Mahajan C. Postoperative Cognitive Dysfunction. Indian J Crit Care Med. 2019 Jun;23(Suppl 2):S162-S164. doi: 10.5005/jp-journals-10071-23196. PMID 31485127
- [Background] Fournier A, Krause R, Winterer G, Schneider R. Biomarkers of postoperative delirium and cognitive dysfunction. Front Aging Neurosci. 2015 Jun 9;7:112. doi: 10.3389/fnagi.2015.00112. eCollection 2015. PMID 26106326
- [Background] Li RL, Zhang ZZ, Peng M, Wu Y, Zhang JJ, Wang CY, Wang YL. Postoperative impairment of cognitive function in old mice: a possible role for neuroinflammation mediated by HMGB1, S100B, and RAGE. J Surg Res. 2013 Dec;185(2):815-24. doi: 10.1016/j.jss.2013.06.043. Epub 2013 Jul 17. PMID 23899512